CLINICAL TRIAL: NCT02053740
Title: Use of Traditional Chinese Medicine (Ren Shen Yang Rong Tang) Against Microinflammation in Hemodialysis Patients: A Quasi-randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Po-Jen Hsiao, Department of Nephrology, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TSGH 2012-1
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Immune Dysfunction
MeSH Terms: conditions — Immune System Diseases | interventions — WW Domain-Containing Oxidoreductase

ARMS (2):
- R-S-Y-R-T (Experimental): We added R-S-Y-R-T (500 mg 3 times per day) for 6 months
  Interventions: Drug: Add R-S-Y-R-T (500 mg 3 times per day) for 6 months; Drug: Routine western medicine
- Routine western medicine (Other): We kept routine western medicine only (as control group)
  Interventions: Drug: Routine western medicine

INTERVENTIONS:
Drug: Add R-S-Y-R-T (500 mg 3 times per day) for 6 months
  Arms: R-S-Y-R-T
Drug: Routine western medicine

SUMMARY:
Participants and study design:

Subjects were recruited and selected for uremic patients on maintenance hemodialysis (HD) who informed us of their interest in the investigators study and were mentally capable to give an informed written consent and willing to comply with study requirements. The inclusion criteria were 18 years or older, with at least 3 months maintenance HD. The exclusion criteria were malignancy, acute infection, gastrointestinal bleeding, pregnancy, and inability to comply with the requirements of study.

69 respondents were enrolled in this trial. A single-center quasi-randomized controlled clinical trial was designed based on the patients in the care of one attending physician. Eligible subjects were allocated to study and control group, and the basic characteristics between the experimental group and control group were matched. There was no significant difference regarding gender, aged, education level, comorbidities between these two groups. The experimental group was treated with Ren Shen Yang Rong Tang (R-S-Y-R-T) combined routine western medicine, and the control group was treated with WM alone. The experimental group had 32 respondents and the control group had 37 respondents. The duration of use of R-S-Y-R-T was 6 months. Finally, there were 27 patients in the experimental group and 32 patients in the control group completed the study. Blood investigation, including biochemical profiles and inflammatory markers were checked at intervals 0, 2, 4 and 6 months form routine HD. The questionnaire, for the assessment of quality of life (QOL) was evaluated at interval 0, and 6 months.

DETAILED DESCRIPTION:
Study medication and dosage:

For this study, the investigators used herbal granules prepared according to the formula of R-S-Y-R-T. The investigators purchased the study products from a manufacturer with a Good Manufacturing Practice (Si Wu Tang) certification in Taiwan. This was a concentrated decoction made by water extraction in 1:13 ratio from single batched roots of the 14 plants in proportions: Radix Paeoniae alba (Bai Sau) (90 g), Radix Angelicae sinensis (Dang Guay) (30 g), Pericarpium Citri Reticulatae (Chenpi) (30 g), Radix Astragali (Huangqi) (30 g), Cortex Cinnamomi (Rougui) (30 g), Radix Ginseng (Renshen) (30 g), Rhizoma Atractylodis Macrocephalae (Baizhu) (30 g), Radix Glycyrrhizae (Gancao) (30 g), Radix Rehmanniae praeparata (Soe Dee Huang) (20 g), Fructus Schisandrae (Wuweizi) (20 g), Poria cocos (Fuling) (20 g), Cortex et Radix Polygalae (Yuanzhi) (15 g), Zingiber officinale Roscoe (Jiang) (30 g)，Fructus Jujubae (Dazao) (10 g) as prepared according to the original pharmacopoeia. The plant origins in China were known to the buyer of the pharmaceutical company and the final product was free of E. coli, Salmonella and pesticide residues. The levels of heavy metals were 1.238 ppm for lead, 0.228 ppm for arsenic,0.10 ppm for cadmium, and <0.0022 ppm for mercury, all within regulated limits (5, 5, 0.5, and 0.5 ppm, respectively). Each pack weighed approximately 500 mg in aluminum packets.

The investigators determined the dosage of 1 pack a time for 3 times a day with warm water for 6 months. The exact number of packs taken was recorded in clinic visits and any unfinished packs were brought back to the study nurse at the next clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years or older
* With maintenance HD for at least 3 months

Exclusion Criteria:

* Malignancy
* Acute infection
* Gastrointestinal bleeding
* Pregnancy
* Inability to comply with the requirements of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | Average 26 weeks (6 months)
  These inflammatory markers include c-reactive protein (CRP), interleukin-6 (IL-6), and tumor necrosis factor-α (TNF-α). We use the xMAP serum assay for the 3 cytokines.

SECONDARY OUTCOMES:
Quality of life | Average 26 weeks (6 months)
  We use the Taiwan version of the WHOQOL-BREF (WHOQOL-BREF [TW]).

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service general hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Background] Nakai S, Kawakita T, Nagasawa H, Himeno K, Nomoto K. Thymus-dependent effects of a traditional Chinese medicine, ren-shen-yang-rong-tang (Japanese name; Ninjin-youei-to), in autoimmune MRI/MP-lpr/lpr mice. Int J Immunopharmacol. 1996 Apr;18(4):271-9. doi: 10.1016/0192-0561(96)84507-3. PMID 8894807
- [Background] Harigai E, Nakai S, Kawakita T, Nomoto K. Combined treatment with ren-shen-yang-rong-tang (Japanese name: ninjin-youei-to) plus prednisolone on adjuvant-induced arthritis in Lewis rat. Int J Immunopharmacol. 1995 May;17(5):411-8. doi: 10.1016/0192-0561(95)00018-w. PMID 7591365
- [Background] Aoki T, Kojima T, Kameda N, Yoshijima S, Ono A, Kobayashi Y. [Anti-inflammatory effect of a traditional Chinese medicine, ren-shen-yang-rong-tang (Japanese name: ninjin-youei-to), on alveolar macrophages stimulated by RANTES or TNF-alpha]. Arerugi. 1994 May;43(5):663-7. Japanese. PMID 7518231